CLINICAL TRIAL: NCT01332136
Title: Determinants of Medical and Surgical Treatment Outcomes in Chronic Sinusitis
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Dr. Timothy L. Smith, Professor, Oregon Health and Science University
Other Study IDs: 2R01DC005805 (NIH)
Record Dates: First submitted 2011-04-07; First posted 2011-04-08 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Rhinosinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sinonasal mucosal tissue specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Endoscopic sinus surgery: Patients electing endoscopic sinus surgery for chronic rhinosinusitis
- Medical management: Continued medical management for symptoms of chronic rhinosinusitis

SUMMARY:
This research study will be completed by enrolling a prospective, observational cohort study to evaluate medical versus surgical treatment outcomes for chronic sinus disease. This investigation will compare quality of life outcomes between each treatment type, as well as measure cellular and molecular markers of inflammation in the sinus mucosa, to create models that predict improvement in quality of life following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>= 18 years)
* Chronic rhinosinusitis as defined by the 2007 multi-disciplinary adult sinusitis guidelines
* Able to complete all surveys/questionnaires in English
* Persistent symptoms following initial medical management
* Received at least 1 course of broad spectrum antibiotics or culture directed antibiotics for at least a total of 14 days
* Received at least a 3 week trial of topical steroid sprays OR at least a 5 day trial of systemic corticosteroid therapy.
* Counseled for subsequent treatment options including either medical management or endoscopic sinus surgery

Exclusion Criteria:

* Children (<18 years)
* Unable to complete all surveys/questionnaires at baseline

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have failed intial medical management for chronic sinusitis and have presented to a tertiary care clinic for continued treatment.
Sampling Method: Non-Probability Sample
Enrollment: 966 (Actual)
Dates: Start 2011-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Disease-specific quality of life | 18 months post-treatment

SECONDARY OUTCOMES:
General health-related quality-of-life | 18 months post-treatment
Olfaction | 18 months post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Patel PA, Kallenberger EM, Nguyen SA, Mace JC, Duffy AN, Soler ZM, Smith TL, Schlosser RJ. Factors Affecting Nasal Discharge in Chronic Rhinosinusitis Patients. Laryngoscope. 2025 Nov;135(11):4086-4092. doi: 10.1002/lary.32288. Epub 2025 May 26. PMID 40417805
- [Derived] Ramakrishnan VR, Arbet J, Mace JC, Suresh K, Shintani Smith S, Soler ZM, Smith TL. Predicting olfactory loss in chronic rhinosinusitis using machine learning. Chem Senses. 2021 Jan 1;46:bjab042. doi: 10.1093/chemse/bjab042. PMID 34473227
- [Derived] Soudry E, Mace J, Smith TL, Hwang PH. Role of inferior turbinate reduction in the quality of life of patients undergoing endoscopic sinus surgery for chronic rhinosinusitis. Int Forum Allergy Rhinol. 2019 Aug;9(8):926-933. doi: 10.1002/alr.22356. Epub 2019 Jun 20. PMID 31220413
- [Derived] Ramakrishnan VR, Mace JC, Soler ZM, Smith TL. Is greater antibiotic therapy prior to ESS associated with differences in surgical outcomes in CRS? Laryngoscope. 2019 Mar;129(3):558-566. doi: 10.1002/lary.27651. Epub 2018 Dec 24. PMID 30582166
- [Derived] Chowdhury NI, Mace JC, Bodner TE, Alt JA, Deconde AS, Levy JM, Smith TL. Does Medical Therapy Improve SinoNasal Outcomes Test-22 Domain Scores? An Analysis of Clinically Important Differences. Laryngoscope. 2019 Jan;129(1):31-36. doi: 10.1002/lary.27470. Epub 2018 Sep 12. PMID 30208209
- [Derived] Beswick DM, Mace JC, Soler ZM, Ayoub NF, Rudmik L, DeConde AS, Smith TL. Appropriateness criteria predict outcomes for sinus surgery and may aid in future patient selection. Laryngoscope. 2018 Nov;128(11):2448-2454. doi: 10.1002/lary.27227. Epub 2018 May 14. PMID 29756211
- [Derived] Error M, Ashby S, Orlandi RR, Alt JA. Single-Blinded Prospective Implementation of a Preoperative Imaging Checklist for Endoscopic Sinus Surgery. Otolaryngol Head Neck Surg. 2018 Jan;158(1):177-180. doi: 10.1177/0194599817731740. Epub 2017 Sep 19. PMID 28925320
- [Derived] DeConde AS, Mace JC, Ramakrishnan VR, Alt JA, Smith TL. Analysis of factors associated with electing endoscopic sinus surgery. Laryngoscope. 2018 Feb;128(2):304-310. doi: 10.1002/lary.26788. Epub 2017 Aug 4. PMID 28776718
- [Derived] Ramakrishnan VR, Mace JC, Soler ZM, Smith TL. Examination of high-antibiotic users in a multi-institutional cohort of chronic rhinosinusitis patients. Int Forum Allergy Rhinol. 2017 Apr;7(4):343-351. doi: 10.1002/alr.21903. Epub 2017 Jan 13. PMID 28084683
- [Derived] DeConde AS, Mace JC, Levy JM, Rudmik L, Alt JA, Smith TL. Prevalence of polyp recurrence after endoscopic sinus surgery for chronic rhinosinusitis with nasal polyposis. Laryngoscope. 2017 Mar;127(3):550-555. doi: 10.1002/lary.26391. Epub 2016 Nov 12. PMID 27859303
- [Derived] Steele TO, Buniel MC, Mace JC, El Rassi E, Smith TL. Lymphoma of the nasal cavity and paranasal sinuses: A case series. Am J Rhinol Allergy. 2016 Sep;30(5):335-9. doi: 10.2500/ajra.2016.30.4347. PMID 27657899
- [Derived] Levy JM, Rudmik L, Peters AT, Wise SK, Rotenberg BW, Smith TL. Contemporary management of chronic rhinosinusitis with nasal polyposis in aspirin-exacerbated respiratory disease: an evidence-based review with recommendations. Int Forum Allergy Rhinol. 2016 Dec;6(12):1273-1283. doi: 10.1002/alr.21826. Epub 2016 Aug 2. PMID 27480830
- [Derived] Falco JJ, Thomas AJ, Quin X, Ashby S, Mace JC, Deconde AS, Smith TL, Alt JA. Lack of correlation between patient reported location and severity of facial pain and radiographic burden of disease in chronic rhinosinusitis. Int Forum Allergy Rhinol. 2016 Nov;6(11):1173-1181. doi: 10.1002/alr.21797. Epub 2016 Jul 20. PMID 27438938
- [Derived] Levy JM, Mace JC, Rudmik L, Soler ZM, Smith TL. Low 22-item sinonasal outcome test scores in chronic rhinosinusitis: Why do patients seek treatment? Laryngoscope. 2017 Jan;127(1):22-28. doi: 10.1002/lary.26157. Epub 2016 Jul 5. PMID 27377575
- [Derived] Steele TO, Mace JC, Dedhia R, Rudmik L, Smith TL, Alt JA. Health utility values for patients with recurrent acute rhinosinusitis undergoing endoscopic sinus surgery: a nested case control study. Int Forum Allergy Rhinol. 2016 Nov;6(11):1182-1187. doi: 10.1002/alr.21809. Epub 2016 Jun 16. PMID 27309906
- [Derived] Smith TL, Mace JC, Rudmik L, Schlosser RJ, Hwang PH, Alt JA, Soler ZM. Comparing surgeon outcomes in endoscopic sinus surgery for chronic rhinosinusitis. Laryngoscope. 2017 Jan;127(1):14-21. doi: 10.1002/lary.26095. Epub 2016 Jun 14. PMID 27298069
- [Derived] Levy JM, Mace JC, Sansoni ER, Soler ZM, Smith TL. Longitudinal improvement and stability of olfactory function in the evaluation of surgical management for chronic rhinosinusitis. Int Forum Allergy Rhinol. 2016 Nov;6(11):1188-1195. doi: 10.1002/alr.21800. Epub 2016 May 24. PMID 27218483
- [Derived] Levy JM, Mace JC, DeConde AS, Steele TO, Smith TL. Improvements in psychological dysfunction after endoscopic sinus surgery for patients with chronic rhinosinusitis. Int Forum Allergy Rhinol. 2016 Sep;6(9):906-13. doi: 10.1002/alr.21776. Epub 2016 Apr 15. PMID 27080574
- [Derived] Cox DR, Ashby S, DeConde AS, Mace JC, Orlandi RR, Smith TL, Alt JA. Dyad of pain and depression in chronic rhinosinusitis. Int Forum Allergy Rhinol. 2016 Mar;6(3):308-14. doi: 10.1002/alr.21664. Epub 2015 Nov 19. PMID 26954903
- [Derived] Abuzeid WM, Mace JC, Costa ML, Rudmik L, Soler ZM, Kim GS, Smith TL, Hwang PH. Outcomes of chronic frontal sinusitis treated with ethmoidectomy: a prospective study. Int Forum Allergy Rhinol. 2016 Jun;6(6):597-604. doi: 10.1002/alr.21726. Epub 2016 Feb 16. PMID 26879467
- [Derived] Steele TO, Rudmik L, Mace JC, DeConde AS, Alt JA, Smith TL. Patient-centered decision making: the role of the baseline SNOT-22 in predicting outcomes for medical management of chronic rhinosinusitis. Int Forum Allergy Rhinol. 2016 Jun;6(6):590-6. doi: 10.1002/alr.21721. Epub 2016 Feb 8. PMID 26852743
- [Derived] Soler ZM, Hyer JM, Rudmik L, Ramakrishnan V, Smith TL, Schlosser RJ. Cluster analysis and prediction of treatment outcomes for chronic rhinosinusitis. J Allergy Clin Immunol. 2016 Apr;137(4):1054-1062. doi: 10.1016/j.jaci.2015.11.019. Epub 2016 Jan 22. PMID 26806047
- [Derived] Steele TO, Detwiller KY, Mace JC, Strong EB, Smith TL, Alt JA. Productivity outcomes following endoscopic sinus surgery for recurrent acute rhinosinusitis. Laryngoscope. 2016 May;126(5):1046-53. doi: 10.1002/lary.25705. Epub 2016 Jan 9. PMID 26749066
- [Derived] DeConde AS, Bodner TE, Mace JC, Alt JA, Rudmik L, Smith TL. Development of a clinically relevant endoscopic grading system for chronic rhinosinusitis using canonical correlation analysis. Int Forum Allergy Rhinol. 2016 May;6(5):478-85. doi: 10.1002/alr.21683. Epub 2015 Dec 17. PMID 26678860
- [Derived] El Rassi E, Mace JC, Steele TO, Alt JA, Smith TL. Improvements in sleep-related symptoms after endoscopic sinus surgery in patients with chronic rhinosinusitis. Int Forum Allergy Rhinol. 2016 Apr;6(4):414-22. doi: 10.1002/alr.21682. Epub 2015 Dec 17. PMID 26678684
- [Derived] El Rassi E, Mace JC, Steele TO, Alt JA, Soler ZM, Fu R, Smith TL. Sensitivity analysis and diagnostic accuracy of the Brief Smell Identification Test in patients with chronic rhinosinusitis. Int Forum Allergy Rhinol. 2016 Mar;6(3):287-92. doi: 10.1002/alr.21670. Epub 2015 Dec 1. PMID 26625169
- [Derived] Alt JA, DeConde AS, Mace JC, Steele TO, Orlandi RR, Smith TL. Quality of Life in Patients With Chronic Rhinosinusitis and Sleep Dysfunction Undergoing Endoscopic Sinus Surgery: A Pilot Investigation of Comorbid Obstructive Sleep Apnea. JAMA Otolaryngol Head Neck Surg. 2015 Oct;141(10):873-81. doi: 10.1001/jamaoto.2015.1673. PMID 26356240
- [Derived] Tarasidis GS, DeConde AS, Mace JC, Ashby S, Smith TL, Orlandi RR, Alt JA. Cognitive dysfunction associated with pain and quality of life in chronic rhinosinusitis. Int Forum Allergy Rhinol. 2015 Nov;5(11):1004-9. doi: 10.1002/alr.21578. Epub 2015 Jun 22. PMID 26246436
- [Derived] Luk LJ, Steele TO, Mace JC, Soler ZM, Rudmik L, Smith TL. Health utility outcomes in patients undergoing medical management for chronic rhinosinusitis: a prospective multiinstitutional study. Int Forum Allergy Rhinol. 2015 Nov;5(11):1018-27. doi: 10.1002/alr.21588. Epub 2015 Jul 3. PMID 26140502
- [Derived] DeConde AS, Mace JC, Ashby S, Smith TL, Orlandi RR, Alt JA. Characterization of facial pain associated with chronic rhinosinusitis using validated pain evaluation instruments. Int Forum Allergy Rhinol. 2015 Aug;5(8):682-90. doi: 10.1002/alr.21539. Epub 2015 Jun 13. PMID 26074476
- [Derived] Soler ZM, Pallanch JF, Sansoni ER, Jones CS, Lawrence LA, Schlosser RJ, Mace JC, Smith TL. Volumetric computed tomography analysis of the olfactory cleft in patients with chronic rhinosinusitis. Int Forum Allergy Rhinol. 2015 Sep;5(9):846-54. doi: 10.1002/alr.21552. Epub 2015 May 26. PMID 26010298
- [Derived] Steele TO, Mace JC, Smith TL. Does comorbid anxiety predict quality of life outcomes in patients with chronic rhinosinusitis following endoscopic sinus surgery? Int Forum Allergy Rhinol. 2015 Sep;5(9):829-38. doi: 10.1002/alr.21543. Epub 2015 Apr 23. PMID 25908106
- [Derived] Sansoni ER, Sautter NB, Mace JC, Smith TL, Yawn JR, Lawrence LA, Schlosser RJ, Soler ZM, Mulligan JK. Vitamin D3 as a novel regulator of basic fibroblast growth factor in chronic rhinosinusitis with nasal polyposis. Int Forum Allergy Rhinol. 2015 Mar;5(3):191-6. doi: 10.1002/alr.21474. Epub 2015 Jan 5. PMID 25561293
- [Derived] DeConde AS, Mace JC, Alt JA, Rudmik L, Soler ZM, Smith TL. Longitudinal improvement and stability of the SNOT-22 survey in the evaluation of surgical management for chronic rhinosinusitis. Int Forum Allergy Rhinol. 2015 Mar;5(3):233-9. doi: 10.1002/alr.21458. Epub 2014 Dec 15. PMID 25511442
- [Derived] DeConde AS, Mace JC, Bodner T, Hwang PH, Rudmik L, Soler ZM, Smith TL. SNOT-22 quality of life domains differentially predict treatment modality selection in chronic rhinosinusitis. Int Forum Allergy Rhinol. 2014 Dec;4(12):972-9. doi: 10.1002/alr.21408. Epub 2014 Oct 16. PMID 25323055
- [Derived] DeConde AS, Mace JC, Alt JA, Soler ZM, Orlandi RR, Smith TL. Investigation of change in cardinal symptoms of chronic rhinosinusitis after surgical or ongoing medical management. Int Forum Allergy Rhinol. 2015 Jan;5(1):36-45. doi: 10.1002/alr.21410. Epub 2014 Sep 18. PMID 25236780
- [Derived] DeConde AS, Barton MD, Mace JC, Smith TL. Can sinus anatomy predict quality of life outcomes and operative times of endoscopic frontal sinus surgery? Am J Otolaryngol. 2015 Jan-Feb;36(1):13-9. doi: 10.1016/j.amjoto.2014.08.011. Epub 2014 Aug 27. PMID 25228283
- [Derived] Smith KA, Smith TL, Mace JC, Rudmik L. Endoscopic sinus surgery compared to continued medical therapy for patients with refractory chronic rhinosinusitis. Int Forum Allergy Rhinol. 2014 Oct;4(10):823-7. doi: 10.1002/alr.21366. Epub 2014 Sep 11. PMID 25213088
- [Derived] Detwiller KY, Smith TL, Alt JA, Trune DR, Mace JC, Sautter NB. Differential expression of innate immunity genes in chronic rhinosinusitis. Am J Rhinol Allergy. 2014 Sep-Oct;28(5):374-7. doi: 10.2500/ajra.2014.28.4082. PMID 25198021
- [Derived] DeConde AS, Bodner TE, Mace JC, Smith TL. Response shift in quality of life after endoscopic sinus surgery for chronic rhinosinusitis. JAMA Otolaryngol Head Neck Surg. 2014 Aug;140(8):712-9. doi: 10.1001/jamaoto.2014.1045. PMID 25074504
- [Derived] DeConde AS, Mace JC, Smith TL. The impact of comorbid gastroesophageal reflux disease on endoscopic sinus surgery quality-of-life outcomes. Int Forum Allergy Rhinol. 2014 Aug;4(8):663-9. doi: 10.1002/alr.21333. Epub 2014 Apr 10. PMID 24723428
- [Derived] DeConde AS, Mace JC, Smith TL. The impact of comorbid migraine on quality-of-life outcomes after endoscopic sinus surgery. Laryngoscope. 2014 Aug;124(8):1750-5. doi: 10.1002/lary.24592. Epub 2014 Feb 20. PMID 24431279
- [Derived] Alt JA, Mace JC, Buniel MC, Soler ZM, Smith TL. Predictors of olfactory dysfunction in rhinosinusitis using the brief smell identification test. Laryngoscope. 2014 Jul;124(7):E259-66. doi: 10.1002/lary.24587. Epub 2014 Feb 10. PMID 24402746
- [Derived] Smith KA, Rudmik L. Impact of continued medical therapy in patients with refractory chronic rhinosinusitis. Int Forum Allergy Rhinol. 2014 Jan;4(1):34-8. doi: 10.1002/alr.21238. Epub 2013 Oct 25. PMID 24166890
- [Derived] Alt JA, Sautter NB, Mace JC, Detwiller KY, Smith TL. Antisomnogenic cytokines, quality of life, and chronic rhinosinusitis: a pilot study. Laryngoscope. 2014 Apr;124(4):E107-14. doi: 10.1002/lary.24412. Epub 2013 Oct 22. PMID 24115141
- [Derived] Alt JA, Smith TL. Chronic rhinosinusitis and sleep: a contemporary review. Int Forum Allergy Rhinol. 2013 Nov;3(11):941-9. doi: 10.1002/alr.21217. Epub 2013 Aug 26. PMID 24039230
- [Derived] Alt JA, Smith TL, Mace JC, Soler ZM. Sleep quality and disease severity in patients with chronic rhinosinusitis. Laryngoscope. 2013 Oct;123(10):2364-70. doi: 10.1002/lary.24040. Epub 2013 Aug 5. PMID 23918740
- [Derived] Soler ZM, Rudmik L, Hwang PH, Mace JC, Schlosser RJ, Smith TL. Patient-centered decision making in the treatment of chronic rhinosinusitis. Laryngoscope. 2013 Oct;123(10):2341-6. doi: 10.1002/lary.24027. Epub 2013 Jul 15. PMID 23856802
- [Derived] Henriquez OA, Schlosser RJ, Mace JC, Smith TL, Soler ZM. Impact of synechiae after endoscopic sinus surgery on long-term outcomes in chronic rhinosinusitis. Laryngoscope. 2013 Nov;123(11):2615-9. doi: 10.1002/lary.24150. Epub 2013 May 13. PMID 23670876
- [Derived] Detwiller KY, Smith TL, Mace JC, Trune DR, Sautter NB. Steroid-independent upregulation of matrix metalloproteinase 9 in chronic rhinosinusitis patients with radiographic evidence of osteitis. Int Forum Allergy Rhinol. 2013 May;3(5):364-8. doi: 10.1002/alr.21135. Epub 2013 Feb 8. PMID 23401274